CLINICAL TRIAL: NCT05904080
Title: Randomized Phase 2 Study of Nivolumab and Ipilimumab With or Without Cabozantinib in Patients With Advanced Nasopharyngeal Carcinoma That Have Progressed After Platinum Treatment and Immunotherapy
Brief Title: Testing Nivolumab and Ipilimumab Immunotherapy With or Without the Targeted Drug Cabozantinib in Recurrent, Metastatic, or Incurable Nasopharyngeal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-04469; NCI-2023-04469 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A092105 (Other: Alliance for Clinical Trials in Oncology); A092105 (Other: CTEP); U10CA180821 (NIH); NCT06010095 (obsolete NCT alias)
Record Dates: First submitted 2023-06-13; First posted 2023-06-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Nasopharyngeal Carcinoma; Recurrent Nasopharyngeal Carcinoma; Stage IV Nasopharyngeal Carcinoma AJCC v8
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Specimen Handling; cabozantinib; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (nivolumab, ipilimumab) (Active Comparator): Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab
- Arm B (nivolumab, ipilimumab, cabozantinib) (Experimental): Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1 and cabozantinib S-malate PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients may continue with cabozantinib S-malate after 2 years per treating investigator. Patients undergo CT or MRI and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
  Arms: Arm B (nivolumab, ipilimumab, cabozantinib)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase II trial tests how well nivolumab and ipilimumab immunotherapy with or without cabozantinib works in treating patients with nasopharyngeal cancer that has come back (after a period of improvement) (recurrent), has spread from where it first started (primary site) to other places in the body (metastatic), or for which no treatment is currently available (incurable). Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Cabozantinib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals cancer cells to multiply. This helps slow or stop the spread of cancer cells. Giving immunotherapy with nivolumab and ipilimumab and targeted therapy with cabozantinib may help shrink and stabilize nasopharyngeal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the progression-free survival (PFS) of the triplet combination (cabozantinib S-malate, nivolumab, and ipilimumab [CaboNivoIpi]) is more favorable than the doublet (nivolumab and ipilimumab [NivoIpi]).

SECONDARY OBJECTIVES:

I. To compare safety and tolerability between the two arms (Common Terminology Criteria for Adverse Events [CTCAE] version [v]5.0.).

II. To compare overall response rate (ORR) between the two arms via both Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune-modified Response Evaluation Criteria in Solid Tumors (iRECIST) criteria.

III. To compare overall survival (OS) between the two arms. IV. To assess response by primary or acquired PD-1/L1 inhibitor resistance in the prior line of therapy.

EXPLORATORY OBJECTIVE:

I. To evaluate molecular and immunologic predictors of response (Epstein-Barr virus [EBV] viral load; PD-L1 score) between arms.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive nivolumab intravenously (IV) over 30 minutes and ipilimumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) and collection of blood samples throughout the trial.

ARM B: Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1 and cabozantinib S-malate orally (PO) daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients may continue with cabozantinib S-malate after 2 years per treating investigator. Patients undergo CT or MRI and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up every 8-12 weeks until progression of disease occurs or a new non-protocol anti-cancer therapy is initiated and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented nasopharyngeal carcinoma (NPC) regardless of World Health Organization (WHO) classification (keratinizing squamous cell carcinoma, non-keratinizing, or basaloid squamous cell carcinoma) and regardless of association with Epstein-Barr virus (EBV) and/or human papillomavirus (HPV)
* Recurrent, metastatic and incurable disease treated with platinum-gemcitabine and prior PD-1/L1 blockade (as first or second-line therapy) where immunotherapy was part of the most recent prior line of therapy
* Patients are eligible regardless of prior smoking history, p16 immunohistochemistry (IHC) status, PD-L1 expression status, EBV tumor status, EBV viral load at baseline, or tumor genomic alteration status
* Patients must have at least one measurable lesion (by RECIST v1.1) which has not been previously irradiated that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions as >= 10 mm (>= 1 cm) (and short axis for nodal lesions, LN >= 15 mm) with CT scan, MRI, or calipers by clinical exam
* Patients may have had no more than 2 prior lines of prior systemic therapy for recurrent, metastatic NPC
* No prior VEGFR targeted therapy permitted
* Age >= 18 years
* Eastern Cooperative Oncology Group Performance (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Hemoglobin >= 9 g/dL
* Platelet count >= 100,000/mm^3
* Creatinine or creatinine clearance =< 1.5 mg/dL or >= 30 Modification of Diet in Renal Disease (MDRD)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN); except subjects with Gilbert syndrome who can have a total bilirubin < 3 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGT]) =< 3 x upper limit of normal (ULN)

  * Up to =< 5 allowed with liver metastases
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown. Therefore, for women of childbearing potential only, a negative urine or serum pregnancy test, per institution standard, done =< 7 days prior to registration is required.

  * Pregnant women are excluded from this study because nivolumab, ipilimumab, and cabozantinib are all Class C or D agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants, secondary to treatment of the mother with any of the study agents, breastfeeding should be discontinued if the mother is treated with as part of this study (in either arm)
* No active tumor bleeding: or radiographic evidence of major blood vessel infiltration as judged by the treating investigator
* Prior -anti-cancer therapy is allowed: Patients need to be recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1), with the exception of alopecia. Any life-threatening events clearly attributable to prior immunotherapy exposure that have a high possibility of recurring should warrant exclusion: including severe pneumonitis, grade 4 bullous dermatitis/drug reaction with eosinophilia and systemic symptoms (DRESS), neurologic events such as autoimmune encephalitis transverse myelitis, and/or myocarditis. Maintenance hormonal replacement or long-term hormonal therapy exposure is permitted.

  * No chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to registration. Palliative (limited-field) radiation therapy is permitted, if all of the following criteria are met:

    * Repeat imaging demonstrates no new sites of bone metastases.
    * The lesion being considered for palliative radiation is not a target lesion
* No patients with a prior malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Brain metastases allowed: Patients with treated brain metastases are eligible if follow-up brain imaging 3 weeks after central nervous system (CNS)-directed therapy shows no evidence of progression. Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial
* For patients with evidence of chronic hepatitis B (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated

  * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently receiving treatment, they are eligible if they have an undetectable HCV viral load
* Solid organ or tissue transplant is allowed: - subsequent therapy with nivolumab increases the risk of organ/tissue rejection. Patients must be instructed that it is crucial they stay in touch with their transplant team during treatment
* No active autoimmune disease: or history of autoimmune disease that might recur, and which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. These include but are not limited to patients with a history of

  * Immune related neurologic disease,
  * Multiple sclerosis,
  * Autoimmune (demyelinating) neuropathy,
  * Guillain-Barre syndrome (GBS),
  * Myasthenia gravis;
  * Systemic autoimmune disease such as SLE,
  * Connective tissue diseases,
  * Scleroderma, inflammatory bowel disease (IBD),
  * Crohn's, ulcerative colitis,
  * Patients with a history of toxic epidermal necrolysis (TEN),
  * Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease
* Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible
* Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome, and psoriasis controlled with topical medication and patients with only positive serology, such as antinuclear antibodies (ANA) or anti-thyroid antibodies, should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Pneumonitis should be evaluated for the nature of the disease process, need for treatment prior study treatment, and the risk of exacerbation with study treatment
* Able to swallow oral medication: No known medical condition causing an inability to swallow oral formulations of agents
* No condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study registration. Patients are permitted the use of topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Adrenal replacement steroid doses > 10 mg daily prednisone are permitted. A brief (less than 3 weeks) course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by a contact allergen) is permitted
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel) is prohibited. Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* Concomitant use of any medications or substances that are strong inhibitors or inducers of CYP3A4 is discouraged; if unavoidable, the dose of cabozantinib on study should be adjusted accordingly. Any complementary medications (e.g., herbal supplements or traditional Chinese medicines) intended to treat the disease under study are prohibited

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2028-06-16 (Estimated); Study Completion 2028-06-16 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to the first of either progression or death from any cause, or censored at last known tumor assessment date, assessed up to 2 years
  PFS will be estimated using the Kaplan-Meier method, where the log-rank test will be used to compare the 2 treatment arms.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, or censored at last known follow-up, assessed up to 2 years
  OS will be estimated using the Kaplan-Meier method, where the log-rank test will be used to compare the 2 treatment arms.
Incidence of adverse events | Up to 2 years
  The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events version 5.0. The frequency and percentage of grade 3+ adverse events will be compared between the 2 treatment arms. Comparisons between arms will be made by using either the chi-square or Fisher's exact test.
Response by subgroups of interest | Up to 2 years
  Will also report and compare the overall response rate (ORR) between different subgroups of interest (primary or acquired PD-1/L1 inhibitor resistance in the prior line of therapy (further defined below), etc.). These comparisons will be done via chi-square or Fisher's exact tests. We'll also assess primary versus acquired resistance to prior PD-1 inhibition in each arm as well. While not a formal stratification, in the interim and final analysis we'll also descriptively assess these subgroups between arms as well.
ORR | Up to 2 years
  The response rate will be compared via chi-square or Fisher's exact tests between the 2 treatment arms using both the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria and also separately for the immune-modified RECIST criteria.
Predictors of response | Up to 2 years
  Will correlate the baseline data (Epstein-Barr virus viral load, p16 immunohistochemistry status, smoking history, and PD-L1 score) with ORR data. For this analysis, logistic regression models will be assessed using the baseline data to predict binary response data. Odds ratios and 95% confidence intervals will be reported. Will also summarize the data using descriptive statistics and graphical methods.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Hanna, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (92):
- United States (92):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MEJ, Council Bluffs, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital South, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm